CLINICAL TRIAL: NCT02871622
Title: A Post-market Registry of the BioMatrix Alpha TM (Cobalt Chromium Biolimus A9TM (BA9TM) Drug-eluting Stent)
Brief Title: BMX Alpha Registry: a Post-market Registry of the BioMatrix Alpha TM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Biosensors Europe SA (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: 16EU01
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease; Stable Angina; Ischemia; Acute Coronary Syndrome; NSTEMI; STEMI
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Ischemia; Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: BioMatrix AlphaTM — Cobalt Chromium BA9 TM drug-eluting stent

SUMMARY:
Prospective, multi-center, registry designed to enrol up to 2,000 patients in up to 35 International centers. All patients will receive a BioMatrix AlphaTM stent as per clinical practice and will be followed for 2 years for data collection. Major adverse cardiac events (MACE) results at 9 months will be compared to the results obtained from the BioMatrix FlexTM arm of the LEADERS trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the BioMatrix AlphaTM stent per clinical indication and physician's choice;
* Patients who agree to comply with the follow up requirements;
* Patients with a life expectancy of > 1 year at time of consent;
* Patients eligible to receive dual anti platelet therapy (DAPT) according to guidelines;
* Hemodynamically stable patients.

Exclusion Criteria:

* Inability to provide informed consent;
* Currently participating in another trial before reaching primary endpoint;
* Planned surgery within 6 months of percutaneous coronary intervention (PCI) unless dual antiplatelet therapy is maintained throughout the perisurgical period;
* Patient has received an additional stent different from a BioMatrix AlphaTM stent during the index procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: "Real world, all comers" patient population: Patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) in the overall population, defined as composite of cardiac death, myocardial infarction (Q-wave and non-Q-wave), or clinically driven target vessel revascularization (TVR). | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian BA Menown, Dr, Principal Investigator — Craigavon Cardiac Centre
Locations (1):
- Craigavon Cardiac Center, Craigavon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not planned